CLINICAL TRIAL: NCT05557851
Title: A Phase 1b, Open-Label, Safety, Pharmacokinetic, and Pharmacodynamic Study of an Anti-super-enhancer Minnelide Given Along With Abraxane Plus Gemcitabine in Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Minnelide Along With Abraxane Plus Gemcitabine in Patients With Metastatic Adenocarcinoma of the Pancreas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneamrita Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minnelide_ACP_101
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 14-O-phosphonooxymethyltriptolide disodium salt

STUDY DESIGN:
Intervention Model Description: Stressing the patient's pancreatic cancer by giving the anti super-enhancer MinnelideTM to increase endoplasmic reticulum (ER) stress and improve the progression-free survival (PFS) when patients are treated with standard of care (SOC) nanoparticle albumin-bound (nab)-paclitaxel (Abraxane) plus gemcitabine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Study of Minnelide in Patients with Metastatic Adenocarcinoma of the Pancreas (Experimental): This is an open-label, Phase 1b study of MinnelideTM given once a day on Days 1 to 5, Days 8 to12 and Days 15 to 19 in combination with SOC (nab-paclitaxel [Abraxane] plus gemcitabine). The study will be conducted in patients with disease progression while on FOLFIRINOX as first treatment and who have had no prior treatment with nab-paclitaxel (Abraxane) plus gemcitabine or single agent nab paclitaxel or gemcitabine or in any other combinations. The total number of treatment cycles administered will be dependent on drug tolerability by patient.
  Interventions: Combination Product: Minnelide

INTERVENTIONS:
Combination Product: Minnelide — Stressing the patient's pancreatic cancer by giving the anti super-enhancer Minnelide to increase endoplasmic reticulum (ER) stress and improve the progression-free survival (PFS) when patients are treated with standard of care (SOC) nanoparticle albumin-bound (nab)-paclitaxel (Abraxane) plus gemcitabine.

SUMMARY:
A Phase 1b, Open-Label, Safety, Pharmacokinetic, and Pharmacodynamic Study of an Anti-super-enhancer Minnelide Once a Day on Days 1 to 5, Days 8 to 12 and Days 15 to 19 Along with Abraxane Plus Gemcitabine in Patients with Metastatic Adenocarcinoma of the Pancreas

DETAILED DESCRIPTION:
Stressing the patient's pancreatic cancer by giving the anti-super-enhancer Minnelide to increase endoplasmic reticulum (ER) stress and improve the progression-free survival (PFS) when patients are treated with standard of care (SOC) nanoparticle albumin-bound (nab)-paclitaxel (Abraxane) plus gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* • Signed, written IRB-approved informed consent.

  * Patients diagnosed with histologically confirmed metastatic adenocarcinoma of the pancreas combined with adenocarcinoma and adenosquamous are allowed, but pure adenosquamous patients are excluded.
  * Disease progression while on FOLFIRINOX as first treatment.
  * Had no prior treatment with nab-paclitaxel (Abraxane) plus gemcitabine or single agent nab-paclitaxel or gemcitabine or in any other combinations.
  * Patient who has received prior or going to receive any killed vaccine including influenza, pneumococcal or COVID-19 during the study are allowed but any live vaccine like Herpes Zoster is not allowed. One or more metastatic tumours measurable on computed tomography (CT) scan per Response Evaluation Criteria in Solid Tumours (RECIST) V1.1 criteria excluding the primary pancreatic lesion.
  * Karnofsky performance ≥ 70%.
  * Life expectancy of at least 3 months, as determined by the Investigator.
  * Age ≥ 19 years.
  * A negative pregnancy test (if female).
  * Acceptable liver function as per below:

    * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
    * Aspartate aminotransferase (AST), serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT), serum glutamic pyruvic transaminase (SGPT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN (if liver metastases are present, then ≤ 5 × ULN is allowed).
    * Albumin ≥ 3.0 g/dL.
  * Acceptable renal function as per below:

    o Serum creatinine within normal limits, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * Acceptable haematologic status:

    * Baseline absolute neutrophil counts ≥ 2000 cells/mm3.
    * Platelet count ≥ 100000 cells/mm3.
    * Haemoglobin ≥ 9 g/dL.
  * Urinalysis: No clinically significant abnormalities.
  * Acceptable coagulation status in the absence of therapeutic intent to anticoagulate:

    * Prothrombin time (PT) ≤ 1.5 × institutional ULN.
    * Partial thromboplastin time (PTT) ≤ 1.5 × institutional ULN.
    * International normalised ratio (INR) ≤ 1.5 × institutional ULN. Note: Abnormal lab values will be retested once within 2 weeks.
  * For men and women of childbearing potential, the use of effective contraceptive methods during the study. From last dose effective contraception is to be maintained as follows:

    * Men: 100 days from last dose of MinnelideTM.
    * Women of childbearing potential: 6 months from last dose of MinnelideTM.
  * For females, agree to the use of two physician-approved contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomised partner) while on study IP, and for 3 months following the last dose of IP.
  * Has negative serum pregnancy test (β-hCG) result at Screening.
  * For males, must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* • New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischaemia on ECG.

  * Baseline QTc exceeding 470 msec (using the Bazett's formula) and/or patients receiving class 1A or class III antiarrhythmic agents. Note: If a single value of QTcB> 470 msec is observed which is not clinically significant as per the Investigator, triplicate ECGs should be performed and if the average QTcB ≤ 470 msec, then the patient can be included in the study.
  * Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
  * Pregnant or nursing women. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her PI immediately.
  * Treatment with radiation therapy (local therapy, non target lesion within 2 weeks), major surgery, chemotherapy, biological agents, or investigational therapy within 3 weeks prior to study treatment.
  * Unwillingness or inability to comply with procedures required in this protocol.
  * Known infection with HIV, hepatitis B, or hepatitis C except for chronic hepatitis B or C patients with undetectable viral load.
  * Serious non-malignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
  * Any other malignancy within 5 years prior to study drug administration, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, or non-melanomatous skin cancer (all treatment of which should have been completed 6 months prior to enrollment).
  * Patient with a history or current evidence of brain metastasis or leptomeningeal disease.
  * Currently receiving any other investigational agent.
  * On a prohibited medication (clarithromycin, loperamide, ondansetron, poly (ADP) - ribose polymerase inhibitors, programmed cell death protein 1 inhibitors, and tyrosine kinase inhibitors or immunotherapeutics).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of Minnelide capsules when given in combination with SOC | 24 months
  To observe any increase in the number of patients that experience Grade 4 neutropenia lasting ≥ 5 days or Grade 3 or 4 neutropenia with fever and/or infection; Grade 4 thrombocytopenia (or Grade 3 with bleeding); Grade 3 or 4 treatment-related non-hematological toxicity (Grade 3 nausea, vomiting or diarrhea that last > 72 hours despite maximal treatment when Minnelide is given in combination of gemcitabine and nab-paclitaxel compared to the incidence with gemcitabine and nab-paclitaxel.

SECONDARY OUTCOMES:
pharmacokinetics of Minnelide and to determine the pharmacodynamics of GRP78 | 24 months
  To determine the pharmacokinetics of Minnelide when given in combination with gemcitabine and nab-paclitaxel
  Plasma concentration data will be used to determine the following PK parameters:
  * AUC Area under the concentration curve
  * Cmax Maximum plasma concentration
  * Tmax Time to maximum plasma concentration
  * t1/2 Terminal phase half life
  * CL/F Total body clearance
  * Vd/F Apparent volume of distribution
  * To determine the effects of Minnelide on the pharmacodynamics of GRP78

CONTACTS AND LOCATIONS:
Overall Officials: Joon Oh Park, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Soeul, South Korea

IPD SHARING:
Plan to Share IPD: No